CLINICAL TRIAL: NCT01506622
Title: Comparison Between Propofol and Fentanyl for Prevention of Emergence Agitation in Children After Sevoflurane Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 4-2010-0536
Record Dates: First submitted 2011-12-25; First posted 2012-01-10 (Estimated); Last update posted 2015-07-16 (Estimated); Status verified 2015-07

CONDITIONS: Emergence Agitation
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Propofol group (Active Comparator): intravenous administration of propofol 1 mg/kg at the end of anesthesia
  Interventions: Drug: Administration of propofol
- Fentanyl group (Active Comparator): intravenous administration of fentanyl 1 mcg/kg at the end of anesthesia
  Interventions: Drug: Administration of fentanyl
- Control group (Active Comparator): intravenous administration of saline at the end of anesthesia
  Interventions: Drug: Administration of saline

INTERVENTIONS:
Drug: Administration of propofol — Propofol 1 mg/kg will be administered to propofol group at the end of anesthesia.
  Arms: Propofol group
Drug: Administration of fentanyl — Fentanyl 1 mcg/kg will be administered to fentanyl group at the end of anesthesia.
  Arms: Fentanyl group
Drug: Administration of saline — Saline will be administered to control group at the end of anesthesia.
  Arms: Control group

SUMMARY:
The occurrence of emergence agitation (EA) in pediatric patients who have received sevoflurane anesthesia is a common postoperative problem. The prevalence of EA varies between 10% to 80% depending on the scoring system for evaluation and the anesthetic technique used.

Many authors reported various strategies such as use of sedative premedication, change of maintenance technique of anesthesia, or pharmacological agents administered at the end of anesthesia to reduce the incidence and severity of EA, and to allow a smooth emergence from sevoflurane anesthesia. Among these strategies, the use of pharmacological agents at the end of anesthesia is not affected by anesthetic duration, and may not prolong recovery duration of anesthesia excessively when these agents are administered as subhypnotic or small dose. The typical agents that can be administered in this way are propofol and fentanyl.

Previous studies demonstrated that the use of either propofol or fentanyl at the end of anesthesia could reduce the incidence of EA.

The purpose of this study is to compare the preventive effect on EA and the characteristics of anesthesia recovery between propofol and fentanyl administered at the end of sevoflurane anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists I or II,
* 18-72 months of age,
* scheduled for ambulatory inguinal hernia repair undergoing general sevoflurane anesthesia

Exclusion Criteria:

* developmental delay
* psychological and neurologic disorder
* sedatives medication
* an abnormal airway
* reactive airway disease
* extreme agitation and uncooperation
* previous history of anesthesia

Ages: 18 Months to 72 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 222 (Actual)
Dates: Start 2011-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
The incidence of emergence agitation | Participants will be followed for the duration of postanesthesia care unit (PACU) stay, an expected average of one hour.
  The investigator will evaluate the incidence and extent of emergence agitation of participants, according to Aono's scale, the 5-step Emergence Agitation (EA) scale. Also, the Pediatric Anesthesia Emergence Delirium (PAED) scale will be used to assess emergence agitation. Aono's scale scores ≥3, 5-step (EA) scale ≥4 or PAED scale scores ≥10 will be considered as presence of emergence agitation

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei University, Seoul, South Korea

REFERENCES:
- [Background] Chen J, Li W, Hu X, Wang D. Emergence agitation after cataract surgery in children: a comparison of midazolam, propofol and ketamine. Paediatr Anaesth. 2010 Sep;20(9):873-9. doi: 10.1111/j.1460-9592.2010.03375.x. PMID 20716081